CLINICAL TRIAL: NCT06899295
Title: Data from Advanced Respiratory Monitoring During Alveolar Recruitment Maneuvers (ARM). a Prospective Observational Study
Brief Title: Prevention of Postoperative Respiratory Complications
Acronym: RAMAGE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: M3DISIM (Other); INSERM UMR-942, Paris, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241304; 2024-A01853-44 (Other: IDRCB)
Record Dates: First submitted 2025-02-24; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: General Anesthesia; Ventilator-Induced Lung Injuries; Postoperative Respiratory Complications
Keywords: Ventilator optimization; Ventilator induced lung injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury | interventions — Hemodynamics; Temperature; Sex; Body Height; Body Mass Index; Laparoscopy; Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Continuous measurement of esophageal pressure Peso (cmH2O) — This parameter will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia.
Diagnostic Test: Measurement of impedance variation with each respiratory cycle (EIT), Z in ohm — This parameter will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia
Diagnostic Test: Measurement of regional respiratory compliance (EIT), Ohm/cmH2O — This parameter will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia
Diagnostic Test: Measurement of lung volumes (EELV or CRF) mL, (ml/kg) — These parameters will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia
Diagnostic Test: Continuous measurement of multiparametric monitoring data in place (hemodynamics, depth of sedation, respiratory data, temperature). — These parameters will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia
Diagnostic Test: Quantification of delivered doses of hypnotics, morphine and paralytics — These parameters will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia
Diagnostic Test: Demographic criteria: age, sex, height, weight, BMI, theoretical ideal weight, ASA. - Procedure-related criteria: type of surgery, technique (laparoscopic, endoscopic, laparoscopic), position, duratio — These parameters will be recorded during the perioperative hospitalization

SUMMARY:
Given the huge number of patients mechanically ventilated during general anaesthesia, optimizing alveolar recruitment by limiting pulmonary and systemic aggression is a key objective for further progress in perioperative patient management.

During general anaesthesia, ventilation disorders with atelectasis, derecruitment of posteroinferior zones and reduced functional residual capacity (FRC) occur in relation to the operative position, the effect of neuromuscular block and general anaesthesia. These conditions of poor pulmonary aeration favor postoperative respiratory complications and are responsible for excess mortality in the perioperative period.

Alveolar recruitment maneuvers (ARMs) are ventilatory strategies used during general anesthesia that aim to restore lung aeration with Positive End Expiratory Pressure (PEEP) sufficient to keep the lungs open afterwards. This pulmonary hyperinflation not only has a major impact on hemodynamics but also presents a risk of barotrauma. ARM is currently performed without precise measurement of the pressures prevailing in the lung.

Advanced monitoring is now available and integrated into the latest-generation ventilators and includes the combination of Transpulmonary pressure (TPP) and Electro-Impedance Tomography " (EIT) measurements.

The aim of this observational study is to measure and record advanced respiratory monitoring data in a minimally invasive way, during alveolar recruitment tests routinely performed for the target population (obese, prone, laparoscopic surgery). Describe and a posteriori analyze the recorded data and establish a relationship between the PEEP values set by conventional ARM and those determined by advanced monitoring combining EIT and PTP for the same patient.

DETAILED DESCRIPTION:
During general anaesthesia, ventilation disorders with atelectasis, derecruitment of posteroinferior zones and reduced functional residual capacity (FRC) occur in relation to the operative position, the effect of neuromuscular block and general anaesthesia. These conditions of poor pulmonary aeration favor postoperative respiratory complications and are responsible for excess mortality in the perioperative period.

Alveolar recruitment maneuvers (ARMs) are ventilatory strategies used during general anesthesia that aim to restore lung aeration with a Positive End Expiratory Pressure (PEEP) sufficient to keep the lungs open afterwards. These maneuvers can be performed in a variety of ways but generally involve gradually increasing the level of airway pressure, followed by a stepwise decrease to an end-expiratory pressure (PEEP) level decided by the practitioner based on monitoring data and considering the clinical outcome and hemodynamic tolerance of the maneuver.

Atelectasis essentially occurs when the pressure in the alveolus at the end of expiration is lower than the pressure that allows the alveolus to remain open (critical opening pressure). The principle is to transiently increase transpulmonary pressure (TTP) (the difference between airway pressure (Paw) and pleural pressure) above the critical opening pressure.

Maintaining alveolar end-expiratory pressure (PEEP) after the maneuver is essential to avoid de-recruitment. The concept of the alveolar recruitment maneuver is very popular in our specialty. The benefits and importance of this alveolar recruitment strategy were initially identified in intensive care patients. Particular attention is now being paid to lung-free patients in the operating theatre, especially those with obesity, during long prone surgeries and during laparoscopic abdominal surgery. Currently, the benefits of ARM are also being seen, with a reduced risk of serious pulmonary and extra-pulmonary complications in the first 7 days postoperatively for this type of patient.

Currently, these maneuvers are performed directly on ventilators that incorporate an automated, programmable procedure. The technique consists in gradually increasing inspiratory pressure to 40 cmH2O and PEEP to 20 cmH2O, the incremental phase. As soon as the maximum pressure level is reached, a progressive decrement phase follows. Three parameters need to be set: maximum inspiratory pressure, maximum PEEP and maneuver duration. The level of PEEP at which the alveoli theoretically remain open is determined by monitoring the patient's compliance and tidal volume. This pulmonary hyperinflation not only has a major impact on hemodynamics but also presents a risk of barotrauma. ARM is currently performed without transpulmonary pressure measurement and with this procedure.

For this reason, new-generation ventilators are equipped with an esophageal pressure proxy for pleural pressure, enabling precise calculation of transpulmonary pressure. Only direct measurement of the parameters characterizing the state of the entire respiratory system enables individual, patient-specific adjustment of the critical opening pressure of the alveoli.

Advanced monitoring is now available and integrated into the latest-generation ventilators, and includes the following combination of measurements obtained from the monitors:

1. Ventilator-integrated

   * Transpulmonary pressure (TPP) is defined as the difference between airway pressure and pleural pressure and provides essential information for individual patient needs on chest wall mechanics, lung mechanics and effects on the respiratory and circulatory systems. Estimation of trans-pulmonary pressure (TPP), pulmonary stress and critical opening pressure is obtained via esophageal manometry (proxy for pleural pressure), the use of which is recommended by several learned societies and is the subject of numerous studies.
   * The study of lung volumes (end-expiratory lung volume, EELV, and a substitute for functional respiratory capacity (FRC) via the study of exhaled CO2 kinetics (volumetric capnography and dynamic capnometry).
2. Electro-Impedance Tomography (EIT) Electro-Impedance Tomography (EIT) provides a totally non-invasive, cross-sectional visualization of part of the pulmonary aeration, both dynamically and regionally. Current technology also enables us to assess pulmonary perfusion (and thus ventilation/perfusion ratios).

Advantages of this augmented and integrative respiratory monitoring approach during mechanical ventilation under general anesthesia:

1. Limiting pulmonary stress, excessive and individualizing the setting of tidal volume (TV) and positive end-expiratory pressure (PEEP) to optimize the acceptable recruitment/distension balance.
2. Obtain information on the gas exchanger and the impact of PEEP-VT optimization on gas exchange.

These maneuvers, with their risk of alveolar overdistension, are potentially dangerous for patients with airway pathologies or difficult ventilator adaptation conditions.

Consequently, the practice of applying a fixed standardized maneuver to a particular patient is risky, and more rigorous control of the optimal end-expiratory pressure level PEEP (critical opening pressure) from advanced monitoring data would be desirable. Customization of this alveolar recruitment maneuver is particularly suited to the population we will be studying (obese, prone, laparoscopic surgery).

The application of MRA during anesthesia normalizes pulmonary function intraoperatively. There is physiological evidence that patients of all ages, whatever the type of surgery, benefit from such active intervention. The risks must be minimized.

The aim of this observational study is to measure and record advanced respiratory monitoring data in a minimally invasive way, during alveolar recruitment tests routinely performed for the target population (obese, prone, laparoscopic surgery). To combine data on ventilation/perfusion ratios measured by EIT with optimization of the aeric ventilatory side. Describe and analyze the recorded data a posteriori and establish a relationship between the PEEP values set by conventional ARM and those determined from advanced monitoring combining EIT and TPP. These analyses will enable us to assess the complementarity and added value of these values in practice, and the respective usefulness of the different indices.

Given the enormous volume of patients mechanically ventilated during general anesthesia, optimizing alveolar recruitment by limiting pulmonary and systemic aggression is a key objective for further progress in perioperative patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. undergoing :

   * scheduled surgery at Hospital Lariboisière.
   * scheduled to last more than 2 hours under general anesthesia for abdominal surgery under laparoscopy or surgery in the prone position, or for obese patients with a BMI >35.
   * And for whom the ventilator used includes advanced monitoring
   * for whom placement of a gastric tube is indicated either because of the duration of the procedure or because it is necessary for the surgery.
3. Patient informed and expressing non-opposition to participation in this study

Exclusion Criteria:

* - Patients under 18 years of age.
* Contraindications to esophageal tube placement
* Contraindications to ARMs
* Patient opposed to protocol participation
* Pregnant, parturient or breast-feeding women
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing planned surgery under prolonged general anesthesia (> 2 hour forecast)
  * in prone position Or
  * laparoscopic abdominal surgery Or
  * Obese patients BMI > 35
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Compare the PEEP setting values obtained from a standardized ARM with the theoretical values obtained from advanced monitoring for the same patient. | These parameters will be recorded during the alveolar recruitment maneuvers routinely performed during general anesthesia (one day)
  PEEP levels (cmH2O)

SECONDARY OUTCOMES:
To establish the relationship between the characteristics and combination of monitoring data and the occurrence of postoperative respiratory complications during the 5 postoperative days. | Acquisition and recording of monitoring data and postoperative respiratory complications during the 5 postoperative days (5 days).
  Arozullah score (Risk of postoperative pulmonary complications Arozullah)
Stratify physiological data according to the main phenotypes which determine respiratory mechanics (obesity, prone position, laparoscopic surgery). | Acquisition and recording of monitoring data and postoperative respiratory complications during the 5 postoperative days.
  Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care Paris, France, 75010, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided